CLINICAL TRIAL: NCT04301583
Title: Procyanidin B2 Enriched Cocoa Effects on Mitochondrial Biogenesis
Acronym: PROMETHEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Mar Larrosa, Tenure Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UEM004
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Athletes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sachets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procyanidin B2 enriched cocoa (Active Comparator): Participants receiving cocoa capsules
  Interventions: Dietary Supplement: procyanidin B2 enriched cocoa
- Placebo group (Placebo Comparator): Participants maltodextrin capsules
  Interventions: Dietary Supplement: procyanidin B2 enriched cocoa

INTERVENTIONS:
Dietary Supplement: procyanidin B2 enriched cocoa — Volunteers will intake 5 grams per day of dietary supplement for 10 weeks

SUMMARY:
The purpose of this study is to test how cocoa-rich procyanidin B2 affect the mitochondrial exercise adaptations.

ELIGIBILITY:
Inclusion Criteria:

* Men/Women
* Age between 18 and 45 years
* Aerobic power of oxygen consumption greater than or equal to 55 mL / kg / min

Exclusion Criteria:

* Smoke
* Any chronic disease
* Intake of nutritional or ergogenic supplements
* Chronic medication
* Cocoa allergy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Difference in mitochondrial number | 10 weeks
  Number of mitochondria in blood cells measured by qPCR using mitochondrial COX1 gene and beta globin as housekeeping nuclear gene
Difference in exercise performance | 10 weeks
  Maximum oxygen consumption
  * of incomplete pulmonary gas exchange on VO2 max - Powers - Citado por 318
  * determination of cardiorespiratory fitness and training … - Clark - Citado por 180 Maximum oxygen consumption

CONTACTS AND LOCATIONS:
Overall Officials: Mar Larrosa, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available